CLINICAL TRIAL: NCT06415370
Title: Examining the Relationship Between Home-Delivered Healthy Meals to Seniors and Social Connectedness: A Mixed Methods Study
Brief Title: Food and Friends: Healthy Meals Delivered to You
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Humana Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-0190
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Mental Health Issue; Food Insecurity
Keywords: Food Insecurity; Mental Health; Seniors
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HDHM and Social Interaction (Intervention) (Experimental): Home delivered healthy meals are delivered in-person, including a "friendly visit" with the participant if the participant desires. Student companions will also contact participants at least one time weekly for telephone reassurance and to provide resource referrals.
  Interventions: Behavioral: Home Delivered Healthy Meals; Behavioral: In-person "friendly visits"; Behavioral: Student Companion calls
- HDHM Only (Control) (Experimental): Home delivered healthy meals are delivered directly to the participant or dropped off at the participant's home in a cooler at their front door if they are not available. Any interaction will be limited.
  Interventions: Behavioral: Home Delivered Healthy Meals

INTERVENTIONS:
Behavioral: Home Delivered Healthy Meals — In-person delivery of HDHM at least one time weekly for 12 weeks.
Behavioral: In-person "friendly visits" — "Friendly visits" last approximately 5-10 minutes and include brief "wellness check" questions such as, "How are you doing today?" "Did you try [HDHM recipe] yesterday- how did it taste? Any suggestions for future flavors?" "What are some of the things you plan to do in the next few days?" "Is there anything else you want to share with me?"
  Arms: HDHM and Social Interaction (Intervention)
Behavioral: Student Companion calls — Student Companions call participants at least one time weekly to provide telephone reassurance- i.e., checking on the participant's well-being. These calls may also include referrals to appropriate resources such as NCCARE 360 (statewide network that connects individuals with complex health and social needs, to community resources and service)
  Arms: HDHM and Social Interaction (Intervention)

SUMMARY:
The goal of this clinical trial is to learn if home delivered healthy meals (HDHM) with or without (intervention vs. control) social interaction can impact mental health and food security in adults aged 65 and older who live alone and have trouble accessing food.

The main questions it aims to answer are:

Does HDHM with or without social interaction change the quality of participant food intake? Does HDHM with or without social interaction change the loneliness that participants may experience? Does HDHM with or without social interaction change the depression that participants may experience?

Researchers will compare a group that receives HDHM only to a group that receives HDHM and social interaction to see if there is a difference between the two groups in their experienced loneliness and depression, and the quality of food that they eat.

Participants will receive 12 weeks' worth of HDHM delivered to their home. Half of the participants will receive weekly phone calls from volunteer student "companions) Participants will also be asked to complete questionnaires over the phone at three timepoints (baseline, 6 weeks, and 12 weeks) during the study. Some participants may also be asked to give their opinions on the program via a telephone conversation.

DETAILED DESCRIPTION:
This study is a randomized control trial (RCT) to measure the impact of a combined social interaction and culturally tailored home delivered healthy meals (HDHM) intervention on participants' mental health and food insecurity compared to those in the control group receiving HDHM alone. In addition, the study aims to test the feasibility of including structured, consistent social interactions as part of HDHM.

This study will include a sample size of 60 participants. Participants in the study will be randomized to a HDHM only group (control), or HDHM with social interactions group (intervention). All participants will receive HDHM (a frozen meal product based on the Mediterranean Diet adapted for United States Southeastern taste preferences) for 12 weeks.

The study team will collect data from participants at baseline, 6 weeks, and 12 weeks via a telephone-administered survey.

A subgroup of 10 participants (5 from the intervention, 5 from the control group) will participate in informant interviews to assess feasibility.

ELIGIBILITY:
Inclusion Criteria:

* 65 and older
* Live alone
* Screen positive for food insecurity or have a medical professional concerned about their food security
* Diagnosed with at least 1 diet-related chronic illness
* Be a Medicaid/Medicare dual beneficiary
* Speak English
* Have a microwave

Exclusion Criteria:

* Diagnosis of dementia/Alzheimer's
* Presence of illness or allergies that would preclude consuming HDHM

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Mean Change in Adult Food Security Score | Baseline up to week 12
  Food security status will be assessed using the United States Adult Food Security Survey Module- a 10-item measure that assesses a person's ability to access food. Questions include topics such as having enough food in the house, running out of food due to lack of money, skipping meals, and reducing portion sizes. Scoring range is from 0-10. A higher score represents a lower food security status. Assessed at baseline, week 6, and week 12.
Median Change of Adult Food Security Score | Baseline up to week 12
  Food security status will be assessed using the United States Adult Food Security Survey Module- a 10-item measure that assesses a person's ability to access food. Questions include topics such as having enough food in the house, running out of food due to lack of money, skipping meals, and reducing portion sizes. Scoring range is from 0-10. A higher score represents a lower food security status. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Fruit Eaten Per Day | Baseline up to week 12
  Total cups of fruit eaten per day will be assessed using question 1 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("On average, how many total cups (use your fist as a measure of a cup) of fruit do you eat each day? Count all that you eat whether in a combination dish or by itself"). Scoring range is categorical, with the following answer choices: 0; ½; 1; 1 ½ ; 2; 2 ½; 3; 3 ½; 4 or more. A higher score represents a greater amount of fruit consumed. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Fruit Eaten Per Day | Baseline up to week 12
  Total cups of fruit eaten per day will be assessed using question 1 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("On average, how many total cups (use your fist as a measure of a cup) of fruit do you eat each day? Count all that you eat whether in a combination dish or by itself"). Scoring range is categorical, with the following answer choices: 0; ½; 1; 1 ½ ; 2; 2 ½; 3; 3 ½; 4 or more. A higher score represents a greater amount of fruit consumed. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Vegetables Eaten Per Day | Baseline up to week 12
  Total cups of vegetables eaten per day will be assessed using question 2 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("On average, how many total cups (use your fist as a measure of a cup) of vegetables do you eat each day? Count all that you eat whether in a combination dish or by itself"). Scoring range is categorical, with the following answer choices: 0; ½; 1; 1 ½ ; 2; 2 ½; 3; 3 ½; 4 or more. A higher score represents a greater amount of vegetables consumed. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Vegetables Eaten Per Day | Baseline up to week 12
  Total cups of vegetables eaten per day will be assessed using question 2 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("On average, how many total cups (use your fist as a measure of a cup) of vegetables do you eat each day? Count all that you eat whether in a combination dish or by itself"). Scoring range is categorical, with the following answer choices: 0; ½; 1; 1 ½ ; 2; 2 ½; 3; 3 ½; 4 or more. A higher score represents a greater amount of vegetables consumed. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Water Consumed Per Day | Baseline up to week 12
  Frequency of water consumed per day will be assessed using question 3 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you drink water (count tap, bottled, or sparkling water)?"). Scoring range is from 0-4. A higher score represents a greater frequency of water consumption. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Water Consumed Per Day | Baseline up to week 12
  Frequency of water consumed per day will be assessed using question 3 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you drink water (count tap, bottled, or sparkling water)?"). Scoring range is from 0-4. A higher score represents a greater frequency of water consumption. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Soda Consumed Per Day | Baseline up to week 12
  Frequency of soda consumed per day will be assessed using question 4 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you drink regular (not diet) soda?"). Scoring range is from 0-4. A higher score represents a greater frequency of soda consumption. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Soda Consumed Per Day | Baseline up to week 12
  Frequency of soda consumed per day will be assessed using question 4 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you drink regular (not diet) soda?"). Scoring range is from 0-4. A higher score represents a greater frequency of soda consumption. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Usage of 1% Milk, Skim Milk, and/or Low-fat Yogurt Per Day | Baseline up to week 12
  Usage of 1% milk, skim milk, and/or low-fat yogurt per day will be assessed using question 5 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you use 1% milk, skim milk, and/or low-fat yogurt?"). Scoring range is from 0-4. A higher score represents a greater usage of 1% milk, skim milk, and/or low-fat yogurt. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Usage of 1% Milk, Skim Milk, and/or Low-fat Yogurt Per Day | Baseline up to week 12
  Usage of 1% milk, skim milk, and/or low-fat yogurt per day will be assessed using question 5 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you use 1% milk, skim milk, and/or low-fat yogurt?"). Scoring range is from 0-4. A higher score represents a greater usage of 1% milk, skim milk, and/or low-fat yogurt. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Consumption of Greater Than 1 Kind of Fruit Per Day | Baseline up to week 12
  Frequency of consumption of greater than 1 kind of fruit per day will be assessed using question 6 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("Do you eat more than one kind of fruit each day (apple, peach, berries, etc.)"). Scoring range is from 0-4. A higher score represents a greater frequency of consuming more than one fruit per day. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Consumption of Greater Than 1 Kind of Fruit Per Day | Baseline up to week 12
  Frequency of consumption of greater than 1 kind of fruit per day will be assessed using question 6 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("Do you eat more than one kind of fruit each day (apple, peach, berries, etc.)"). Scoring range is from 0-4. A higher score represents a greater frequency of consuming more than one fruit per day. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Consumption of Greater Than 1 Kind of Vegetable Per Day | Baseline up to week 12
  Frequency of consumption of greater than 1 kind of vegetable per day will be assessed using question 7 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you eat more than one kind of vegetable each day (carrots, corn, green beans, etc.)"). Scoring range is from 0-4. A higher score represents a greater frequency of consuming more than one vegetable per day. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Consumption of Greater Than 1 Kind of Vegetable Per Day (Baseline to Week 6) | Baseline up to week 12
  Frequency of consumption of greater than 1 kind of vegetable per day will be assessed using question 7 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you eat more than one kind of vegetable each day (carrots, corn, green beans, etc.)"). Scoring range is from 0-4. A higher score represents a greater frequency of consuming more than one vegetable per day. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Healthy Food Option Consideration | Baseline up to week 12
  How often someone considers healthy food choices when deciding what to eat will be assessed using question 8 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("When deciding what to eat, how often do you think about healthy food choices?"). Scoring range is from 0-4. A higher score represents a greater frequency considering healthy food choices when deciding what to eat. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Healthy Food Option Consideration | Baseline up to week 12
  How often someone considers healthy food choices when deciding what to eat will be assessed using question 8 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("When deciding what to eat, how often do you think about healthy food choices?"). Scoring range is from 0-4. A higher score represents a greater frequency considering healthy food choices when deciding what to eat. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Usage of "Nutrition Facts" Label | Baseline up to week 12
  How often someone uses a "Nutrition Facts" label to when making food choices will be assessed using question 9 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you use the "Nutrition Facts" on the food label to make food choices?"). Scoring range is from 0-4. A higher score represents a greater frequency of using the "Nutrition Facts" when making food choices. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Usage of "Nutrition Facts" Label | Baseline up to week 12
  How often someone uses a "Nutrition Facts" label to when making food choices will be assessed using question 9 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you use the "Nutrition Facts" on the food label to make food choices?"). Scoring range is from 0-4. A higher score represents a greater frequency of using the "Nutrition Facts" when making food choices. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Consideration of Food Label (Salt/Sodium) | Baseline up to week 12
  How often someone uses a food label to select food with less salt or sodium will be assessed using question 10 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you read food labels to select foods with less salt or sodium?"). Scoring range is from 0-4. A higher score represents a greater frequency of using the food label when making food choices with less salt or sodium. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Consideration of Food Label (Salt/Sodium) | Baseline up to week 12
  How often someone uses a food label to select food with less salt or sodium will be assessed using question 10 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you read food labels to select foods with less salt or sodium?"). Scoring range is from 0-4. A higher score represents a greater frequency of using the food label when making food choices with less salt or sodium. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Consideration of Food Label (Sugar) | Baseline up to week 12
  How often someone uses a food label to select food with less or no added sugar will be assessed using question 11 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you read food labels to select foods with less or no added sugar?"). Scoring range is from 0-4. A higher score represents a greater frequency of using the food label when making food choices with less or no added sugar. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Consideration of Food Label (Sugar) | Baseline up to week 12
  How often someone uses a food label to select food with less or no added sugar will be assessed using question 11 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you read food labels to select foods with less or no added sugar?"). Scoring range is from 0-4. A higher score represents a greater frequency of using the food label when making food choices with less or no added sugar. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Consideration of Food Label (Fat) | Baseline up to week 12
  How often someone uses a food label to select food with less saturated fat will be assessed using question 12 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you read food labels to select foods with less saturated fat?"). Scoring range is from 0-4. A higher score represents a greater frequency of using the food label when making food choices with less saturated fat. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Consideration of Food Label (Fat) | Baseline up to week 12
  How often someone uses a food label to select food with less saturated fat will be assessed using question 12 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you read food labels to select foods with less saturated fat?"). Scoring range is from 0-4. A higher score represents a greater frequency of using the food label when making food choices with less saturated fat. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Whole Grain Consumption | Baseline up to week 12
  How often someone consumes whole grain instead of white or enriched flour ones will be assessed using question 13 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you eat whole grains (whole wheat bread, whole wheat tortillas, brown rice, oatmeal, etc.) in place of white or enriched flour ones?"). Scoring range is from 0-4. A higher score represents a greater frequency of consuming whole grains instead of white or enriched flour ones. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Whole Grain Consumption | Baseline up to week 12
  How often someone consumes whole grain instead of white or enriched flour ones will be assessed using question 13 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How often do you eat whole grains (whole wheat bread, whole wheat tortillas, brown rice, oatmeal, etc.) in place of white or enriched flour ones?"). Scoring range is from 0-4. A higher score represents a greater frequency of consuming whole grains instead of white or enriched flour ones. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Meal Preparation | Baseline up to week 12
  How often someone prepares meals at home will be assessed using question 14 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("Do you prepare meals at home?"). Scoring range is from 0-4. A higher score represents a greater frequency of preparing meals at home. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Meal Preparation | Baseline up to week 12
  How often someone prepares meals at home will be assessed using question 14 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("Do you prepare meals at home?"). Scoring range is from 0-4. A higher score represents a greater frequency of preparing meals at home. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Strength Training | Baseline up to week 12
  How often someone includes strength training when they exercise will be assessed using question 19 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("Do you include strength training when you exercise?"). Scoring range is from 0-4. A higher score represents a greater frequency of strength training. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Strength Training | Baseline up to week 12
  How often someone includes strength training when they exercise will be assessed using question 19 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("Do you include strength training when you exercise?"). Scoring range is from 0-4. A higher score represents a greater frequency of strength training. Assessed at baseline, week 6, and week 12.
Mean Change in Food Frequency Assessment- Physical Activity | Baseline up to week 12
  Participants' amount of physical activity will be assessed using question 20 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How much physical activity (exercise) do you do in a day?"). Scoring is categorical, with the following answer choices: 0-20 minutes; 21-30 minutes; 31-40 minutes; 41-60 minutes; more than 60 minutes. A higher score represents a greater amount of physical activity. Assessed at baseline, week 6, and week 12.
Median Change in Food Frequency Assessment- Physical Activity | Baseline up to week 12
  Participants' amount of physical activity will be assessed using question 20 of a food frequency assessment adapted from the 17-item National Cancer Institute fruit and vegetable screener and the National Health and Nutrition Examination Survey (NHANES) Dietary Screener ("How much physical activity (exercise) do you do in a day?"). Scoring is categorical, with the following answer choices: 0-20 minutes; 21-30 minutes; 31-40 minutes; 41-60 minutes; more than 60 minutes. A higher score represents a greater amount of physical activity. Assessed at baseline, week 6, and week 12.
Mean Change of PRAPARE Score | Baseline up to week 12
  Distinct social determinant of health risks will be assessed using the Protocol for Responding to and Assessing Patients' Assets, Risks, and Experience (PRAPARE) assessment- a 21-item measure that assesses a participant's various social determinant of health risk responses. Questions include topics such as housing status, work situations, level of education, and others. Scoring range is from 0-22, with a higher score representing a higher amount of risks present. Assessed at baseline, week 6, and week 12.
Median Change of PRAPARE Score | Baseline up to week 12
  Distinct social determinant of health risks will be assessed using the Protocol for Responding to and Assessing Patients' Assets, Risks, and Experience (PRAPARE) assessment- a 21-item measure that assesses a participant's various social determinant of health risk responses. Questions include topics such as housing status, work situations, level of education, and others. Scoring range is from 0-22, with a higher score representing a higher amount of risks present. Assessed at baseline, week 6, and week 12.
Mean Change in Patient Health Questionaire-8 | Baseline up to week 12
  Depressive symptoms will be assessed using the Patient Health Questionnaire-8, an 8-item measure that assesses the number of days a person has experienced various symptoms of depression over the past two weeks. Questions include assessing how often a participant has had little to no interest in doing things, how often they feel down, depressed, irritable, or hopeless, etc. Scoring range is from 0-24. A higher score means greater depressive symptoms. Assessed at baseline, week 6, and week 12.
Median Change in Patient Health Questionaire-8 | Baseline up to week 12
  Depressive symptoms will be assessed using the Patient Health Questionnaire-8, an 8-item measure that assesses the number of days a person has experienced various symptoms of depression over the past two weeks. Questions include assessing how often a participant has had little to no interest in doing things, how often they feel down, depressed, irritable, or hopeless, etc. Scoring range is from 0-24. A higher score means greater depressive symptoms. Assessed at baseline, week 6, and week 12.
Mean Change in sum of University of California- Los Angeles Loneliness Scale Short form | Baseline up to week 12
  Loneliness will be assessed using the University of California- Los Angeles Loneliness Scale Short Form, a 6 item measure that assesses how often participants feel left out or not connected to other people. Scoring range is from 3-9. A higher score means greater loneliness. Assessed at baseline, week 6, and week 12.
Median Change in sum of University of California- Los Angeles Loneliness Scale Short form | Baseline up to week 12
  Loneliness will be assessed using the University of California- Los Angeles Loneliness Scale Short Form, a 6 item measure that assesses how often participants feel left out or not connected to other people. Scoring range is from 3-9. A higher score means greater loneliness. Assessed at baseline, week 6, and week 12.
Number of successful HDHM Deliveries made to participants in control group | Baseline up to week 12
  Program feasibility will be assessed using the number of successful HDHM deliveries made to participants during the study. This is defined as the delivery driver being able to deliver the HDHM to the participant's residence. A higher number of successful deliveries indicate greater feasibility.
Number of successful HDHM Deliveries and Social Interactions made to participants in intervention group | Baseline up to week 12
  Program feasibility will be assessed using the number of successful HDHM deliveries including "friendly visits" made to intervention participant's homes during the study. This is defined as the delivery driver being able to deliver the HDHM to the participant's residence and complete a brief social interaction. A higher number of successful deliveries indicates greater feasibility of the program.
Number of HDHM meals consumed by participants weekly | Baseline up to week 12
  Program feasibility will be assessed using the number of meals consumed by participants per week. A higher number of meals consumed indicates greater feasibility of the program.
Duration of Student Companion Calls | Baseline up to week 12
  Program feasibility will be assessed using the duration of Student Companion calls that take place during the study for participants in the intervention group. Duration will be assessed in minutes per week. A higher number of minutes indicates greater feasibility of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Haynes-Maslow, PhD, MHA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.